CLINICAL TRIAL: NCT01202591
Title: A Randomised Double-blind Phase IIa Study (With Combination Safety Run-in) to Assess the Safety and Efficacy of AZD4547 in Combination With Fulvestrant vs. Fulvestrant Alone in ER+ Breast Cancer Patients With FGFR1 Polysomy or Gene Amplification Who Have Progressed Following Treatment With Prior Endocrine Therapy (Adjuvant or First-line Metastatic) (GLOW)
Brief Title: Safety and Efficacy of AZD4547 in Combination With Fulvestrant vs. Fulvestrant Alone in ER+ Breast Cancer Patients
Acronym: GLOW
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D2610C00003; 2010-021220-10 (EudraCT Number)
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-01

CONDITIONS: FGFR Inhibition, Pharmacokinetics, Biomarkers; ER+ Breast Cancer
Keywords: Breast Cancer; ER+; FGFR1; Exemestane; AZD4547; Fulvestrant
MeSH Terms: conditions — Breast Neoplasms | interventions — AZD4547; exemestane; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AZD4547 + exemestane (Experimental): Safety run-in: AZD4547 plus exemestane
  Interventions: Drug: AZD4547; Drug: Exemestane
- AZD4547 + fulvestrant (Experimental): A Randomised phase IIa: AZD4547 plus fulvestrant
  Interventions: Drug: AZD4547; Drug: Fulvestrant
- Placebo + fulvestrant (Placebo Comparator): Randomised phase IIa: Matching placebo plus fulvestrant
  Interventions: Drug: Placebo; Drug: Fulvestrant

INTERVENTIONS:
Drug: AZD4547 — Tablet oral twice daily
  Arms: AZD4547 + exemestane; AZD4547 + fulvestrant
Drug: Exemestane — Tablet oral once daily
  Arms: AZD4547 + exemestane
Drug: Placebo — Tablet oral twice daily
  Arms: Placebo + fulvestrant
Drug: Fulvestrant — A monthly intramuscular injection of a depot formulation with a loading dose 14 days after initial administration
  Arms: AZD4547 + fulvestrant; Placebo + fulvestrant

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of AZD4547 in combination with fulvestrant vs. fulvestrant alone in ER+ breast cancer patients with FGFR1 polysomy (FISH4/5) or gene amplification (FISH 6)

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women (either through bilateral oophorectomy or amenorrhoeic for 24 months)
* Histological confirmation of Breast Cancer with documented ER+ receptor status
* Safety run-in: Relapsing during/within 12 months of completion of a single regimen of adjuvant endocrine therapy with non-steroidal AI and/ tamoxifen or progression following 1st line endocrine therapy with non-steroidal AL
* Rand phase IIa: Received at least 1 prior endocrine therapy in the metastatic setting or have relapsed during/ within 6 months of completion of adjuvant endocrine therapy (either non-steroidal AI or tamoxifen or a combination of both). Chemotherapy administered in the adjuvant setting is permitted.
* Rand phase IIa: Mandatory provision of tumour sample to confirm FGFR1 polysomy or gene amplification. At least one measurable lesion that can be accurately assessed by CT/MRI/x-ray at baseline and follow up visits

Exclusion Criteria:

* Prior exposure to exemestane (safety run-in) / fulvestrant (randomized phase IIa), or any agent known to inhibit FGFRs.
* More than 1 prior regimen of chemotherapy for breast cancer
* ECG recordings that demonstrate significant abnormalities in cardiac rate, rhythm or conduction
* History of hypersensitivity to active or inactive excipients of AZD4547 or exemestane (safety run-in ) or fulvestrant (Randomized phase), including castor oil, or drugs with a similar chemical structure or class to AZD4547 or exemestane or fulvestrant.
* Randomized phase IIa: bleeding/blood clotting conditions that would prevent the administration of the fulvestrant injection into the buttocks

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2010-12; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donal Landers, Study Director — AstraZeneca
Locations (21):
- Belgium (2):
  - Research Site, Leuven
  - Research Site, Namur
- Czechia (2):
  - Research Site, Brno
  - Research Site, Prague
- Research Site, Villejuif, France
- Germany (3):
  - Research Site, Erlangen
  - Research Site, München
  - Research Site, Rostock
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Kaposvár
  - Research Site, Nyíregyháza
  - Research Site, Szeged
- Italy (3):
  - Research Site, Genova
  - Research Site, Lido di Camaiore
  - Research Site, Roma
- Research Site, Cluj-Napoca, Romania
- United Kingdom (5):
  - Research Site, Dundee
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Oxford
  - Research Site, Sutton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient was enrolled on 8 Dec 2010 and Last patient last visit was on 21 Oct 2014. Recruitment was slow, leading to concerns about the feasibility of completing enrolment. Moreover, the limited evidence of clinical activity of AZD4547 monotherapy in FGFR gastric cancer and NSCLC has resulted in a business decision to terminate enrolment.
Pre-assignment Details: Part A: 38 patients enrolled, 31 patients received AZD4547+exemestane; 7 patients did not receive (5 patients were not eligible, 1 patient due to patient decision, 1 patient due to "Other") Part B: 89 patients enrolled; 80 were not eligible, 9 patients received the treatment
Groups:
- AZD4547 80mg bd Cont + Ex 25mg: 80 mg AZD4547 BD continuous + 25 mg exemestane
- AZD4547 40mg Cont + Ex 25mg: 40 mg AZD4547 BD continuous + 25 mg exemestane
- AZD4547 80mg bd 1w/1w + Ex 25mg: 80 mg AZD4547 bd one week on/one week off + 25 mg exemestane
- AZD4547 80mg bd 2w/1w + Ex: 80 mg AZD4547 BD two week on/one week off + 25 mg exemestane
- Part B: AZD4547 + Fulvestrant: 80 mg AZD4547 BD + 500 mg Fulvestrant
- Part B: Placebo + Fulvestrant: 80mg Placebo BD + 500 mg Fulvestrant
Period: Overall Study
Arm/Group | AZD4547 80mg bd Cont + Ex 25mg | AZD4547 40mg Cont + Ex 25mg | AZD4547 80mg bd 1w/1w + Ex 25mg | AZD4547 80mg bd 2w/1w + Ex | Part B: AZD4547 + Fulvestrant | Part B: Placebo + Fulvestrant
Started | 5 | 5 | 12 | 9 | 5 | 4
Completed | 0 | 0 | 1 | 2 | 0 | 0
Not Completed | 5 | 5 | 11 | 7 | 5 | 4
Not completed — Adverse Event | 2 | 1 | 4 | 4 | 0 | 0
Not completed — Other reason as per investigator | 3 | 4 | 7 | 3 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Objective Disease Progression | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- AZD4547 40mg bd Cont + Ex 25mg: 40 mg AZD4547 BD continuous + 25 mg exemestane
- AZD4547 80mg bd 2w/1w + Ex 25mg: 80 mg AZD4547 bd two week on/one week off + 25 mg exemestane
- Part B: Placebo + Fulvestrant: 80 mg Placebo BD + 500 mg Fulvestrant
- Total: Total of all reporting groups
Arm/Group | AZD4547 80mg bd Cont + Ex 25mg | AZD4547 40mg bd Cont + Ex 25mg | AZD4547 80mg bd 1w/1w + Ex 25mg | AZD4547 80mg bd 2w/1w + Ex 25mg | Part B: AZD4547 + Fulvestrant | Part B: Placebo + Fulvestrant | Total
Number analyzed (Participants) | 5 | 5 | 12 | 9 | 5 | 4 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.4 (16.70) [49 to 74] | 61.2 (9.36) [30 to 72] | 66.5 (8.46) [49 to 77] | 67.3 (9.66) [50 to 77] | 61.0 (6.82) | 67.3 (9.46) | 64.6 (10.58) [30 to 77]
Age, Customized [Number; unit: Participants]
  < 35 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  35 >= - < 50 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  50 >= - <65 | 2 | 2 | 3 | 3 | 4 | 1 | 15
  >= 65 | 2 | 2 | 8 | 6 | 1 | 3 | 22
Sex/Gender, Customized [Number; unit: Participants]
  Female | 5 | 5 | 12 | 9 | 5 | 4 | 40
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian (Other Than Chinese And Japanese) | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not Applicable | 2 | 0 | 8 | 4 | 2 | 0 | 16
  Other | 2 | 5 | 4 | 5 | 3 | 4 | 23
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 4 | 5 | 11 | 9 | 5 | 4 | 38
  Other | 1 | 0 | 1 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability in Terms of Number of Patients With Adverse Events (Serious and Non-serious)
Time Frame: 3 years, 10 months (Adverse events recorded from patient screening to discontinuation plus 28 days safety follow-up).
Population: All patients who receive at least one dose of study treatment (AZD4547 or exemestane)
Measure: Number; unit: Participants
Arm/Group | AZD4547 80mg bd Cont + Ex 25mg | AZD4547 40mg Cont + Ex 25mg | AZD4547 80mg bd 1w/1w + Ex 25mg | AZD4547 80mg bd 2w/1w + Ex 25mg | Part B: AZD4547 + Fulvestrant | Part B: Placebo + Fulvestrant
Number analyzed (Participants) | 5 | 5 | 12 | 9 | 5 | 4
Participants | 5 | 5 | 12 | 9 | 5 | 2

ADVERSE EVENTS:
Time Frame: 3 years, 10 months (Adverse events recorded from patient screening to discontinuation plus 28 days safety follow-up).
Arm/Group | AZD4547 80mg bd Cont + Ex 25mg | AZD4547 40mg bd Cont + Ex 25mg | AZD4547 80mg bd 1w/1w + Ex 25mg | AZD4547 80mg bd 2w/1w + Ex 25mg | Part B: AZD4547 + Fulvestrant | Part B: Placebo + Fulvestrant
Serious Adverse Events (participants affected / at risk) | 2/5 | 2/5 | 5/12 | 1/9 | 1/5 | 1/4
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5 | 12/12 | 9/9 | 5/5 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD4547 80mg bd Cont + Ex 25mg (N=5) | AZD4547 40mg bd Cont + Ex 25mg (N=5) | AZD4547 80mg bd 1w/1w + Ex 25mg (N=12) | AZD4547 80mg bd 2w/1w + Ex 25mg (N=9) | Part B: AZD4547 + Fulvestrant (N=5) | Part B: Placebo + Fulvestrant (N=4)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OESOPHAGEAL ACHALASIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEVICE DEPOSIT ISSUE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIC SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLEURAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TROPONIN INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
VIITH NERVE PARALYSIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GAIT DISTURBANCE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE CRISIS OF PSORIASIC OLIGOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | AZD4547 80mg bd Cont + Ex 25mg (N=5) | AZD4547 40mg bd Cont + Ex 25mg (N=5) | AZD4547 80mg bd 1w/1w + Ex 25mg (N=12) | AZD4547 80mg bd 2w/1w + Ex 25mg (N=9) | Part B: AZD4547 + Fulvestrant (N=5) | Part B: Placebo + Fulvestrant (N=4)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHORIORETINOPATHY (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DETACHMENT OF RETINAL PIGMENT EPITHELIUM (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
DRY EYE (Eye disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
EYE DISCHARGE (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE DISORDER (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EYE IRRITATION (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE PAIN (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
EYELID PAIN (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GROWTH OF EYELASHES (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
KERATITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LACRIMATION INCREASED (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
MACULOPATHY (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OCULAR DISCOMFORT (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUBRETINAL FLUID (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ULCERATIVE KERATITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
VISUAL IMPAIRMENT (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VITREOUS FLOATERS (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL MASS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 4 (4) | 4 (4) | 3 (3) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 4 (4) | 3 (3) | 7 (7) | 5 (5) | 4 (4) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FAECAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
GLOSSODYNIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIP DRY (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MELAENA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 5 (5) | 2 (2) | 1 (1)
OESOPHAGEAL SPASM (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PARAESTHESIA ORAL (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 2 (2) | 0 (0)
TONGUE DISCOLOURATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
CRYING (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEVICE BREAKAGE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 3 (3) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
FIBROSIS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INJURY ASSOCIATED WITH DEVICE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOCAL SWELLING (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
CONJUNCTIVITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
GINGIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
LYMPHANGITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MASTITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAIL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
PARONYCHIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION FUNGAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VARICELLA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JOINT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
BLOOD GLUCOSE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLOOD IRON DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD PHOSPHORUS INCREASED (Investigations) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
BODY TEMPERATURE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC ENZYMES INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COLD AGGLUTININS POSITIVE (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM T WAVE ABNORMAL (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INSPIRATORY CAPACITY DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OXYGEN SATURATION DECREASED (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TROPONIN T INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BREAST CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
METASTATIC PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEURILEMMOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AGEUSIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APHASIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 2 (2) | 2 (2) | 6 (6) | 6 (6) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOKINESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
MYOCLONUS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEPRESSED MOOD (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEREALISATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
SLEEP DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BREAST DISORDER (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BREAST PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VULVOVAGINAL DRYNESS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NASAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RALES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINALGIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3) | 6 (6) | 5 (5) | 2 (2) | 0 (0)
BLISTER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 5 (5) | 3 (3) | 2 (2) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
MADAROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NAIL BED BLEEDING (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (4) | 4 (4) | 1 (1) | 0 (0)
NAIL DYSTROPHY (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ONYCHALGIA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ONYCHOLYSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
PAPULE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN HAEMORRHAGE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SWELLING FACE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HOT FLUSH (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LYMPHOEDEMA (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PALLOR (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0/4 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corneal epithelium defect (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post viral fatigue syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrolment to the Part B was terminated on 27 March 2014. Slow recruitment led to concerns that enrolment would not be completed in a realistic timeframe. This led to a business decision to terminate the enrolment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less